CLINICAL TRIAL: NCT00378027
Title: Phase IV, Single Arm Study to Obtain Information Regarding the Safety and Efficacy of Fondaparinux Given Outpatient for Treatment of Acute Pulmonary Embolism
Brief Title: Arixtra PE Study- Outpatient Management of Stable Acute Pulmonary Embolism: Once Daily Subcutaneous Fondaparinux
Status: Withdrawn | Type: Observational
Why Stopped: enrollment criteria not met by PI patient population
Sponsor: The Cleveland Clinic (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 05-202
Record Dates: First submitted 2006-09-18; First posted 2006-09-19 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2017-01

CONDITIONS: Pulmonary Embolism
Keywords: Pulmonary Embolism; PE; Outpatient; Anticoagulation
MeSH Terms: conditions — Pulmonary Embolism | interventions — Fondaparinux

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Stable Acute Pulmonary Embolism: Administer weight dosed Fondaparinux
  Interventions: Drug: Fondaparinux

INTERVENTIONS:
Drug: Fondaparinux — Administer Fondaparinux Risk Stratify
  Other Names: Arixtra

SUMMARY:
To assess the safety and efficacy of outpatient treatment using fondaparinux and oral Vit K antagonist, warfarin (Coumadin) in patients with stable acute pulmonary embolus (APE)when initial therapy is administered in the hospital. Prospectively validate risk stratification criteria for predicting patient suitability for outpatient treatment of acute pulmonary embolism.

DETAILED DESCRIPTION:
The current standard therapy for Acute Pulmonary Embolism (APE) involves admitting patients to the hospital for administration of parenteral anticoagulation therapy(Unfractionated Heparin, Low Molecular Weight Heparin, or Fondaparinux) as a bridge to oral Vitamin K Antagonists (warfarin{Coumadin}). There is a group of patients who are low risk for adverse events and thus may be amenable to outpatient management. Newly identified cardio-specific biomarkers, such as cardiac troponins (TNT and cTnI) and brain natriuretic peptide (BNP) offer added diagnostic information that has been shown to help risk stratify patients presenting with APE. Use of the biomarkers could help separate low- from high-risk subjects, particularly the subgroup of patients who, despite hemodynamic stability at presentation, carry the highest risk of adverse events. Once a low risk APE group is identified, a less complex and less resource-intensive but equally efficacious and safe treatment which allows earlier discharge would be desirable. The current reference therapy is intravenous unfractionated heparin (UFH) for initial anticoagulation for a minimum of 4-5 days of overlap and until therapeutic INR is achieved. Although low-molecular weight heparins (LMWH) have been widely used for DVT treatment, their use for patients with APE is limited to inpatient administration. Fondaparinux sodium (Arixtra) is a synthetic and specific inhibitor of activated Factor X(Xa). Several studies have shown that fondaparinux was more effective than enoxaparin when used as a venous thromboembolism (VTE) prophylaxis agent. Additionally, in the published literature to date, there are no reported cases of heparin-induced thrombocytopenia (HIT) syndrome proven to be caused by fondaparinux. Fondaparinux is approved by the Food and Drug Administration (FDA) for the treatment of acute pulmonary embolism when administered in conjunction with warfarin sodium when initial therapy is administered in the hospital. By means of a non-randomized, open label pilot study, we seek to prospectively assess the safety and efficacy of outpatient treatment using fondaparinux and oral Vitamin K antagonists (warfarin) in patients with stable acute pulmonary embolus and validate risk stratification criteria for predicting patient suitability for outpatient therapy of acute pulmonary embolism.

ELIGIBILITY:
Inclusion Criteria:

Patients enrolled into the trial must meet all of the following criteria:

* At least 18 years of age and able to provide informed consent
* Objectively confirmed symptomatic APE [intraluminal filling defect on spiral computed tomography (CT) or pulmonary angiography, or high- probability ventilation-perfusion (V/Q)lung scan
* Stable and low risk defined as:

  * Hemodynamically stable (HR≤120, no hypotension, no tachypnea, no mental status change, no shock state)
  * O2 supplement ≤4 L/NC
  * Lack of electrocardiographic or echocardiographic evidence for new RV strain
  * Radiographically non-massive PE (absence of saddle emboli on PA gram or spiral CT, perfusion defect on V/Q scan <50%
  * No significant cardiac abnormalities (EF<35%, unstable angina, positive stress test within the past 3 months without revascularization) or pulmonary disease (severe COPD, pulmonary HTN).
  * Negative cardio-specific biomarkers obtained at baseline (TNT, BNP)
  * No moderate or severe RV dysfunction on echocardiogram
* Women of childbearing potential must have a negative pregnancy test (urine or serum) within 24 hours of enrollment

Exclusion Criteria:

Patients meeting one or more of the following criteria are not eligible for enrollment into the trial:

* In the opinion of the clinician, the patient should receive in-patient standard medical therapy
* Contraindication for anticoagulation therapy (active or recent bleeding, recent surgery, bleeding diathesis, recent neurologic event)
* Is receiving therapeutic doses of UFH or LMWH for >24 hours
* Thrombolytic or glycoprotein IIb/IIIa agents administered within 24 hours prior to enrollment
* Platelet count <100,000
* Creatinine clearance <30 mL/min at time of enrollment
* Presence of neuraxial anesthesia and/or post-operative indwelling epidural catheter
* Known history of antiphospholipid antibody syndrome
* Weight >150 kg (330.7 lbs) or <45 kg (99.2 lbs)
* Life expectancy ≤3 months
* Associated arterial thrombosis
* Heparin induced thrombocytopenia (HIT) diagnosed within the past 100 days
* IVC filter
* Any condition that in the opinion of the investigator will prohibit compliance with study procedures and treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stable acute pulmonary embolism
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2006-08 (Actual); Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John R Bartholomew, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic 9500 Euclid Ave., Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Buller HR, Davidson BL, Decousus H, Gallus A, Gent M, Piovella F, Prins MH, Raskob G, van den Berg-Segers AE, Cariou R, Leeuwenkamp O, Lensing AW; Matisse Investigators. Subcutaneous fondaparinux versus intravenous unfractionated heparin in the initial treatment of pulmonary embolism. N Engl J Med. 2003 Oct 30;349(18):1695-702. doi: 10.1056/NEJMoa035451. PMID 14585937